CLINICAL TRIAL: NCT02481869
Title: Does Early Platelet Rich Plasma Injection Decrease the Risk of Post-traumatic Arthritis in Pilon Fractures Undergoing Two-staged Open Reduction With Internal Fixation?
Brief Title: Platelet Rich Plasma Injection in Pilon Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Brett Crist, Assistant Professor, Co-Director of Trauma Services, Co-Director Orthopaedic Trauma Fellowship, Department of Orthopaedic Surgery, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2002117
Record Dates: First submitted 2015-06-11; First posted 2015-06-25 (Estimated); Results first posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-01

CONDITIONS: Fracture
Keywords: Closed; unilateral; pilon
MeSH Terms: conditions — Fractures, Bone | interventions — Arthrocentesis; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arthrocentesis/PRP (Active Comparator): At the time of surgery, the participant will have both injured and uninjured ankles cleaned with surgical soap. An needle will be placed into the injured ankle joint and synovial fluid will be drawn out of the ankle and collected into a syringe. Using the same needle, the PRP will be delivered into the same arthrocentesis needle.
  Next the uninjured ankle will have the same procedure as the injured ankle, except there will be no injection of PRP. There will only be a aspiration of synovial fluid from the uninjured ankle joint using a different clean needle.
  Another aspiration of the synovial fluid will be done at the time of the second surgery in the same manner as before, except there will be no injection of PRP, just an aspiration of both injured and uninjured ankles.
  Interventions: Biological: Arthrocentesis/PRP
- Arthrocentesis/Saline (Placebo Comparator): At the time of surgery, the participant will have both injured and uninjured ankles cleaned with surgical soap. An needle will be placed into the injured ankle joint and synovial fluid will be drawn out of the ankle and collected into a syringe. Using the same needle, the Saline will be delivered into the same arthrocentesis needle.
  Next the uninjured ankle will have the same procedure as the injured ankle, except there will be no injection of Saline. There will only be a aspiration of synovial fluid from the uninjured ankle joint using a different clean needle.
  Another aspiration of the synovial fluid will be done at the time of the second surgery in the same manner as before, except there will be no injection of Saline, just an aspiration of both injured and uninjured ankles.
  Interventions: Drug: Arthrocentesis/Saline

INTERVENTIONS:
Biological: Arthrocentesis/PRP — PRP (n=20): single intra-articular injection of 5 ml of a leukocyte-reduced platelet rich plasma (ACP, Arthrex, Naples, FL) at the time of closed reduction and initial stabilization using ankle-spanning external fixation
  Other Names: platelet-rich plasma
  Arms: Arthrocentesis/PRP
Drug: Arthrocentesis/Saline — Control (n=20): single intra-articular injection of 5 ml of sterile 0.9% saline at the time of closed reduction and initial stabilization using ankle-spanning external fixation
  Other Names: saline
  Arms: Arthrocentesis/Saline

SUMMARY:
Patients who sustain broken ankles have a very high risk of developing arthritis soon after injury (within 2 years). This arthritis can cause increased pain and a decrease level of function, especially if the injury occurs at an early age. During and shortly after ankle injury, there is an inflammatory chemical process that takes place in the ankle that can cause damage to the cartilage in the ankle joint. The investigators want to use what is called Platelet Rich Plasma (PRP), which is produced from a small amount of the patient's own blood, to inject into the injured ankle to see if they can decrease the inflammation that happens after the injury and to see if they can decrease arthritis.

DETAILED DESCRIPTION:
Patients who sustain broken ankles have a very high risk of developing arthritis soon after their injury (within 2 years). This arthritis can cause increased pain and decreased level of function, especially if the injury occurs at an early age. During and shortly after the ankle injury, there is an inflammatory chemical processes that take place in the ankle that can cause damage to the cartilage in the ankle joint. Currently the treatment for this injury is doing surgery is a two step process. When the patient has an ankle fracture, surgeons will stabilize the fracture with an external fixation device to allow ankle swelling to decrease which has been shown improve outcomes within a few hours. After about 10 days the patient will come back for their final surgery in which surgeons will open the ankle joint and make sure that the joint lines up and fix it with plates and screws.

There is no intervention that is done with regards to the physiologic process that goes on inside the ankle joint when the ankle is injured. This is what the investigators intend to study. There is a very large destructive process that may contribute with the early development to arthritis.

The investigators would like to see the effect of this inflammatory response with the addition of platelet rich plasma (PRP) which is produced from a small vial of the patient's own blood. PRP has been used safely in patients with osteoarthritis and has been shown to slow the progression and improve pain scores. PRP is made by spinning the patient's blood in a centrifuge which separates the blood cells from each other. The bloods cells that are anti-inflammatory in nature are taken and placed in another syringe. This is a blinded randomized control study. There will be two groups in which the patients will randomize into: PRP group, or Normal Saline Group. In both groups, the investigator's plan is to withdraw joint fluid from both the injured and uninjured ankle at the time of the first surgery as to analyze the joint fluid from both ankles.

Participants who are randomized into the PRP group will receive PRP in the injured ankle at the time of the first surgery when the external fixator is placed. Participants who are randomized into the Normal Saline group will receive Normal Saline in the injured ankle at the time of the first surgery when the external fixator is placed.

After 7-14 days the participant will return and have their second surgery for definitive fixation. At the time of surgery, joint fluid will again be taken out of the joint for analysis to see if the PRP decreased the anti-inflammatory cells decreased inflammation. After the second surgery the participant will be followed up in the clinic in a regular manner.

ELIGIBILITY:
Inclusion Criteria:

* Closed unilateral pilon fracture

Exclusion Criteria:

* Patients who are younger than 18 years of age
* Open pilon fracture
* Patients with contralateral lower extremity injury
* Patients unable to comply with the follow-up appointments
* Patients who had previous ankle injury to the currently injured ankle
* Patients who are pregnant
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett D Crist, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marsh JL, Weigel DP, Dirschl DR. Tibial plafond fractures. How do these ankles function over time? J Bone Joint Surg Am. 2003 Feb;85(2):287-95. PMID 12571307
- [Background] Martin JA, Buckwalter JA. Post-traumatic osteoarthritis: the role of stress induced chondrocyte damage. Biorheology. 2006;43(3,4):517-21. PMID 16912423
- [Background] Green DM, Noble PC, Ahuero JS, Birdsall HH. Cellular events leading to chondrocyte death after cartilage impact injury. Arthritis Rheum. 2006 May;54(5):1509-17. doi: 10.1002/art.21812. PMID 16649187
- [Background] Guilak F, Fermor B, Keefe FJ, Kraus VB, Olson SA, Pisetsky DS, Setton LA, Weinberg JB. The role of biomechanics and inflammation in cartilage injury and repair. Clin Orthop Relat Res. 2004 Jun;(423):17-26. doi: 10.1097/01.blo.0000131233.83640.91. PMID 15232421
- [Background] Franklin SP, Cook JL. Prospective trial of autologous conditioned plasma versus hyaluronan plus corticosteroid for elbow osteoarthritis in dogs. Can Vet J. 2013 Sep;54(9):881-4. PMID 24155495
- [Background] Waters NP, Stoker AM, Carson WL, Pfeiffer FM, Cook JL. Biomarkers affected by impact velocity and maximum strain of cartilage during injury. J Biomech. 2014 Sep 22;47(12):3185-95. doi: 10.1016/j.jbiomech.2014.06.015. Epub 2014 Jun 21. PMID 25005436
- [Background] Waters NP, Stoker AM, Pfeiffer FM, Cook JL. Biomarkers Affected by Impact Severity during Osteochondral Injury. J Knee Surg. 2015 Jun;28(3):191-200. doi: 10.1055/s-0034-1376329. Epub 2014 May 23. PMID 24858662
- [Background] Garner BC, Stoker AM, Kuroki K, Evans R, Cook CR, Cook JL. Using animal models in osteoarthritis biomarker research. J Knee Surg. 2011 Dec;24(4):251-64. doi: 10.1055/s-0031-1297361. PMID 22303754
- [Background] Thomas TP, Anderson DD, Mosqueda TV, Van Hofwegen CJ, Hillis SL, Marsh JL, Brown TD. Objective CT-based metrics of articular fracture severity to assess risk for posttraumatic osteoarthritis. J Orthop Trauma. 2010 Dec;24(12):764-9. doi: 10.1097/BOT.0b013e3181d7a0aa. PMID 21076249

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Plan for total enrollment of n=40 with n=20 in the PRP arm and n=20 in the saline arm
Groups:
- Platelet Rich Plasma: At the time of surgery, the participant will have both injured and uninjured ankles cleaned with surgical soap. An needle will be placed into the injured ankle joint and synovial fluid will be drawn out of the ankle and collected into a syringe. Using the same needle, the PRP will be delivered into the same arthrocentesis needle.
  Next the uninjured ankle will have the same procedure as the injured ankle, except there will be no injection of PRP. There will only be a aspiration of synovial fluid from the uninjured ankle joint using a different clean needle.
  Another aspiration of the synovial fluid will be done at the time of the second surgery in the same manner as before, except there will be no injection of PRP, just an aspiration of both injured and uninjured ankles.
  Arthrocentesis/PRP: PRP (n=20): single intra-articular injection of 5 ml of a leukocyte-reduced platelet rich plasma (ACP, Arthrex, Naples, FL) at the time of closed reduction and initial stabilization using ankle-s
- Saline: At the time of surgery, the participant will have both injured and uninjured ankles cleaned with surgical soap. An needle will be placed into the injured ankle joint and synovial fluid will be drawn out of the ankle and collected into a syringe. Using the same needle, the Saline will be delivered into the same arthrocentesis needle.
  Next the uninjured ankle will have the same procedure as the injured ankle, except there will be no injection of Saline. There will only be a aspiration of synovial fluid from the uninjured ankle joint using a different clean needle.
  Another aspiration of the synovial fluid will be done at the time of the second surgery in the same manner as before, except there will be no injection of Saline, just an aspiration of both injured and uninjured ankles.
  Arthrocentesis/Saline: Control (n=20): single intra-articular injection of 5 ml of sterile 0.9% saline at the time of closed reduction and initial stabilization using ankle-spanning external fixation
Period: Overall Study
Arm/Group | Platelet Rich Plasma | Saline
Started | 5 | 6
Completed | 0 | 2
Not Completed | 5 | 4
Not completed — Lost to Follow-up | 3 | 4
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Platelet Rich Plasma: At the time of surgery, the participant will have both injured and uninjured ankles cleaned with surgical soap. A needle will be placed into the injured ankle joint and synovial fluid will be drawn out of the ankle and collected. Using the same needle, the PRP will be delivered into the joint.
  Next the uninjured ankle will have the same procedure as the injured ankle, except there will be no injection of PRP. There will only be a aspiration of synovial fluid from the uninjured ankle joint using a different clean needle.
  Another aspiration of the synovial fluid will be done at the time of the second surgery in the same manner as before, except there will be no injection of PRP, just an aspiration of both injured and uninjured ankles.
  Arthrocentesis/PRP: PRP (n=20): single intra-articular injection of 5 ml of a leukocyte-reduced platelet rich plasma (ACP, Arthrex, Naples, FL) at the time of closed reduction and initial stabilization using ankle-spanning external fixation
- Total: Total of all reporting groups
Arm/Group | Platelet Rich Plasma | Saline | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.66 (11.77) | 48.88 (17.97) | 44.47 (15.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Intra-articular Inflammatory Biomarkers at the Time of Definitive Fixation
Description: Inflammatory Biomarkers will be measured (pg/ml) at the time of definitive Fixation
Time Frame: 2 weeks after external fixation
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Platelet Rich Plasma: At the time of surgery, the participant will have both injured and uninjured ankles cleaned with surgical soap. An needle will be placed into the injured ankle joint and synovial fluid will be drawn out of the ankle and collected. Using the same needle, the PRP will be delivered. Next the uninjured ankle will have the same procedure as the injured ankle, except there will be no injection of PRP. There will only be a aspiration of synovial fluid from the uninjured ankle joint using a different clean needle.
  Another aspiration of the synovial fluid will be done at the time of the second surgery in the same manner as before, except there will be no injection of PRP, just an aspiration of both injured and uninjured ankles. Arthrocentesis/PRP: PRP (n=20): single intra-articular injection of 5 ml of a leukocyte-reduced platelet rich plasma (ACP, Arthrex, Naples, FL) at the time of closed reduction and initial stabilization using ankle-spanning external fixation
Arm/Group | Platelet Rich Plasma | Saline
Number analyzed (Participants) | 5 | 6
pg/ml
  Fractaline | 54.89 (44.84) | 163.01 (163.70)
  GRO-A | 2479.17 (1560.321) | 2511.32 (3171.135)
  IL-10 | 37.87 (31.249) | 71.38 (58.70)
  MCP-3 | 109.59 (81.920) | 113.59 (121.850)
  PDGF-AA | 763.67 (770.151) | 284.72 (245.856)
  IL-13 | 0.47 (0.656) | 0.35 (0.341)
  PDGF-ABBB | 3273.77 (2439.361) | 2246.71 (3416.702)
  IL-1RA | 1759.51 (1547.219) | 2690.89 (2015.254)
  IL-1B | 1.62 (1.079) | 5.95 (8.439)
  IL-2 | 0.28 (0.378) | 1.82 (1.756)
  IL-4 | 0.00 (0.000) | 9.08 (20.303)
  IL-6 | 2161.64 (2590.332) | 2206.67 (2584.125)
  IL-8 | 2373.21 (3787.668) | 2554.12 (4199.522)
  MCP-1 | 4290373 (3708.968) | 4152.51 (3541.933)
  MIP-1A | 9.70 (17.591) | 7.44 (5.412)
  MIP-1B | 28.26 (46.006) | 23.11 (10.392)
  TNF-A | 6.21 (2.408) | 6.46 (3.316)
  VEGF | 716.06 (838.759) | 953.47 (1077.999)
  MMP-2 | 49985.40 (24550.313) | 61667.25 (6011.542)
  MMP-1 | 8482.56 (6398.284) | 10643.50 (5011.581)
  MMP-7 | 21182.40 (19303.296) | 43418.25 (37425.332)
  MMP-9 | 23974.72 (36530.879) | 7628.05 (11921.451)
  Prostaglandin E2 (PGE2) | 709.43 (1165.492) | 411.76 (646.284)

2. Primary Outcome: Number of Participants With Presence of Post-traumatic Osteoarthritis 18 Months After Open Reduction Internal Fixation (ORIF)
Description: Post-traumatic Osteoarthritis will be determined from whole-joint Magnetic Resonance Imaging (MRI)
Time Frame: 18 months after ORIF
Population: Only 2 subjects in the Saline group completed the MRI at 18 months after surgery. None of the subjects in the Platelet Rich Plasma (PRP) group completed the MRI
Measure: Count of Participants; unit: Participants
Arm/Group | Platelet Rich Plasma | Saline
Number analyzed (Participants) | 0 | 2
Participants | 0 | 1

3. Secondary Outcome: Patient Reported Outcomes (PROs): Ankle-Hindfoot Scale (AOFAS), Short Form Health Survey (SF-12), and Visual Analog Scale (VAS)
Description: The AOFAS is a standardized evaluation of the clinical status of the ankle-hindfoot. In uses both subjective & objective information. Patients report their pain (40 possible points), physicians assess alignment (10 possible points) & the patient and physician work together to complete the function portion (50 possible points). Total scores range from 0-100, with healthy ankles receiving 100.
  The SF-12 assesses the impact of health on an individual's everyday life. The 2 scores are reported from the SF12 - a mental componet score (MCS) and a physical component score (PCS). The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations (SD). The US average PCS-12 and MCS are both 50 points. The US population SD is 10 points. So each 10 increment of 10 point or above or below 50, corresponds to 1 SD away from the average.
  VAS measures the amount of pain a patient feels on a continuum from 0=no pain to 100=worst pain.
Time Frame: 2 weeks after ORIF
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Platelet Rich Plasma | Saline
Number analyzed (Participants) | 2 | 5
score on a scale
  SF-12 Physical Score | 24.11 (1.95) | 28.96 (4.62)
  SF-12 Mental Score | 58.06 (12.24) | 48.97 (10.47)
  AOFAS Pain Score | 0.00 (0.000) | 6.60 (7.092)
  AOFAS Total Score | 15.00 (21.213) | 15.00 (10.000)
  AOFAS Function Score | 15.00 (21.213) | 19.50 (4.933)
  VAS Score | 5.12 (4.66) | 5.86 (2.87)

4. Secondary Outcome: Patient Reported Outcomes (PROs)
Description: as for outcome 3
Time Frame: 6 weeks after ORIF
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Platelet Rich Plasma | Saline
Number analyzed (Participants) | 2 | 4
score on a scale
  SF-12 Physical Score | 27.47 (11.34) | 34.39 (2.60)
  SF-12 Mental Score | 49.09 (13.16) | 41.48 (5.79)
  AOFAS Pain Score | 15.00 (21.213) | 25.00 (5.774)
  AOFAS Total Score | 15.00 (28.75) | 21.213 (8.808)
  AOFAS Function Score | 0.00 (0.000) | 3.75 (3.775)
  VAS Score | 5.50 (6.36) | 3.33 (1.13)

5. Secondary Outcome: Patient Reported Outcomes (PROs)
Description: as for outcome 3
Time Frame: 12 weeks after ORIF
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Platelet Rich Plasma | Saline
Number analyzed (Participants) | 1 | 4
score on a scale
  SF-12 Physical Score | 37.210 | 42.11 (8.4)
  SF-12 Mental Score | 60.1 | 48.67 (13.24)
  AOFAS Pain Score | 40.00 | 30.00 (8.16)
  AOFAS Total Score | 45.00 | 39.25 (11.383)
  AOFAS Function Score | 5.00 | 9.25 (7.042)
  VAS Score | 1.000 | 1.7625 (1.017)

6. Secondary Outcome: Patient Reported Outcomes (PROs)
Description: as for outcome 3
Time Frame: 6 months after ORIF
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Platelet Rich Plasma | Saline
Number analyzed (Participants) | 1 | 2
score on a scale
  SF-12 Physical Score | 50.62 | 46.54 (8.91)
  SF-12 Mental Score | 61.18 | 39.29 (7.27)
  AOFAS Pain Score | 30.00 | 25.00 (7.071)
  AOFAS Total Score | 45.00 | 39.50 (10.607)
  AOFAS Function Score | 15.00 | 14.50 (3.536)
  VAS Score | 1.000 | 3.87 (2.50)

7. Secondary Outcome: Patient Reported Outcomes (PROs)
Description: as for outcome 3
Time Frame: 12 months after ORIF
Population: Only 2 subjects in the saline group completed the PRO for the 12 months follow up time-frame. All the subjects in the PRP group were lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Platelet Rich Plasma | Saline
Number analyzed (Participants) | 0 | 2
score on a scale
  SF-12 Physical Score |  | 51.14 (5.9)
  SF-12 Mental Score |  | 41.13 (24.88)
  AOFAS Pain Score |  | 30.00 (0.000)
  AOFAS Total Score |  | 46.50 (2.121)
  AOFAS Function Score |  | 16.50 (2.121)
  VAS Score |  | 1.4250 (0.60104)

ADVERSE EVENTS:
Time Frame: 18 months
Description: AEs and SAEs were assessed via a non-systemic approach. Methods of assessment were self-reporting by participants and collection of information from existing medial records for those subjects who did not regularly return for their follow-up visits.
Arm/Group | Platelet Rich Plasma | Saline
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 4/5 | 0/6
Other Adverse Events (participants affected / at risk) | 1/5 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Platelet Rich Plasma (N=5) | Saline (N=6)
Infection (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Hardware Loosening (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Painful Implants (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Painful Implants requiring removal
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Platelet Rich Plasma (N=5) | Saline (N=6)
Post-traumatic Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-08-30): https://cdn.clinicaltrials.gov/large-docs/69/NCT02481869/Prot_000.pdf
  • Statistical Analysis Plan (2016-08-30): https://cdn.clinicaltrials.gov/large-docs/69/NCT02481869/SAP_001.pdf